CLINICAL TRIAL: NCT00431470
Title: Is the Classroom Education Program Intervention Effective in Increasing Positive Self Esteem, Enhancing Leadership Behaviors, While Decreasing the Prevalence of Bullying Behaviors in Fifth Grade Elementary Students?
Brief Title: Are Character Building Lessons Effective in Decreasing Bullying Behaviors?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: M. Governo, Coney Island Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 06/09/VA01
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2006-10

CONDITIONS: Aggression
Keywords: Classroom violence, character, bullying, self esteem
MeSH Terms: conditions — Aggression; Bullying

INTERVENTIONS:
Behavioral: Six classroom based character building education lessons

SUMMARY:
Through the use of an educational intervention, the object of this study is to reduce the prevalence of bullying behaviors among fifth grade school age children. Bullying behaviors promote an environment of violence , fear, and hostility. The study will arrange to present six character education lessons in the classroom of fifth grade students in a New York City public school. Questionnaires will be administered to the students before and after all the lessons have been completed. Questionnaires will collect information about the students self perception of their levels of misconduct, impulsivity, confidence, value of non violence, ways of handling anger, opinions of their leadership behaviors, prevalence of bullying behaviors, and indications of levels of self esteem. Also, their fifth grade teachers will complete pre and post treatment student behavioral questionnaires.

DETAILED DESCRIPTION:
This is a 2 X 2X 2 research design that will study the constructs of self esteem, leadership skills, and prevalence of bullying among a fifth grade school age population. Before data collection, a letter describing the study along with an informed consent sheet, will be mailed to the student's parent/guardian. The written material will state that their child participation is not mandatory. A 48 item likert style questionnaire pre-treatment, post-treatment survey design will be administered to students. Basic demographic questions will also be asked about.

All fifth graders will be given questionnaires before they receive the six classroom lessons of 45 minutes duration and then after all the six lessons have been completed. Lessons will be offered on a weekly basis. The fifth graders will be divided into small groups of approximately 10 individuals. The lessons will be delivered by baccalaureate nursing students in their last semester of college. The groups will be formed at the beginning and membership will remain consistent to enhance development of trust and ease of authentic communication. The lessons will be selected from the program, Overcoming Obstacles, a formal educational program designed to assist students to communicate well and set meaningful goals for their lives. In addition, the classroom teachers will be asked to complete a 14 item likert style pre-treatment, post-treatment, both before and after the six lessons about their opinions of each student's behaviors pattern.

A statistician is a co-investigator and will identify the type of statistical analysis to be done.

ELIGIBILITY:
Inclusion Criteria:

* Fifth grade elementary school students

Exclusion Criteria:

* Special education students

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 175 (Estimated)
Dates: Start 2007-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Questionnaires | Complete

CONTACTS AND LOCATIONS:
Overall Officials: Margaret M Governo, EdD, APRN, Principal Investigator — Coney Island Hospital / Wagner College
Locations (1):
- PS 45, Staten Island, New York, United States